CLINICAL TRIAL: NCT01388413
Title: A Randomized, Multicenter, Parallel Group Study to Evaluate Safety and Efficacy of a Weekly Oral Cyclic Antibiotic Programme in the Prevention of Urinary Tract Infection on Neurological Bladder
Brief Title: Safety and Efficacy of a Weekly Oral Cyclic Antibiotic Programme in the Prevention of Urinary Tract Infection on Neurological Bladder
Acronym: PACHIU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHRI06-LB/PACHIU; 2010-021241-44 (EudraCT Number); A101183-72 (Other: Afssaps); 2010-R31 (Other: CPP)
Record Dates: First submitted 2011-06-23; First posted 2011-07-06 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2017-02

CONDITIONS: Neurogenic Bladder; Urinary Tract Infection
Keywords: neurogenic bladder; urinary tract infection
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly Oral Cyclic Antibiotic programme (Experimental)
  Interventions: Drug: Weekly Oral Cyclic Antibiotic programme
- Classic care (No Intervention)

INTERVENTIONS:
Drug: Weekly Oral Cyclic Antibiotic programme — The Weekly Oral Cyclic Antibiotic Programme consisted of the alternate administration of an antibiotic once per week. The antibiotics that were chosen (efficient for urinary tract infection, well tolerated, low selection pressure) included : Amoxicillin 6000 mg, Amoxicillin/clavulanic acid 3000 mg, Cefixime 400 mg, Fosfomycin trometamol 6000 mg, Trimethoprim/sulfamethoxazole 2400 mg. During week A,the patient received a single antibiotic (A), and the following week B the patient was given another antibiotic (B). For each patient, antibiotics were specifically chosen according to the results of urine cultures.
  Arms: Weekly Oral Cyclic Antibiotic programme

SUMMARY:
Symptomatic urinary tract infections (UTIs) are one of the main causes of morbidity and the main cause of re-hospitalization in subjects with neurogenic bladder. Long-term antibiotic therapy increases the risk of multi-resistant bacterial infections, without reducing the rate of symptomatic UTIs. Our non-comparative preliminary study has shown that Weekly Oral Cyclic Antibiotic Programme (single, weekly dose of antibiotic X on even weeks, and antibiotic Y on odd weeks) seem to drastically reduce both the number of symptomatic UTIs and the number of hospitalizations in patients with neurogenic bladder, without affecting bacterial ecology.

The objective of this study is to validate this preliminary work with a large-scale randomized, parallel-group, multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* subject over 18 years of age
* having a neurogenic bladder with automatic catheter and pharmacologic disconnection of the detrusor muscle
* having at least 4 symptomatic UTIs per year with bacterial sensitivity to the chosen antibiotics
* having given full consent to participate in the study
* being the recipient of social security benefits

Exclusion Criteria:

* known allergy or hypersensitivity to useful antibiotics (to which the bacterium or bacteria are sensitive) or to one of their components
* other contraindication in the administering of useful antibiotics
* urinary volume flow >500 ml during automatic catheter
* different urinary drainage method than automatic catheter
* occurrence of stones in the urinary tract
* infection due to endo urinary material (urinary prosthesis, ureteral stent)
* creatinine clearance <60 ml/min
* patient under guardianship
* women who are pregnant, nursing, or who may become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-08; Primary Completion 2016-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of symptomatic UTIs | During the 6-month follow-up
  Symptomatic UTIs are defined by the presence of infection or reinfection by the same bacteria, in combination with the presence of definite clinical signs of infection (autonomous hyper-reflexivity, spasticity, leakage, contractures, pyuria, fever, shivers).

SECONDARY OUTCOMES:
The number of feverish UTIs | During the 6-month follow-up
  The number of feverish UTIs
The number of hospitalizations | During the 6-month follow-up.
  The number of hospitalizations
The duration of UTI-related hospitalizations | During the 6-month follow-up
  The duration of UTI-related hospitalizations
The tolerance level to the Weekly Oral Cyclic Antibiotic Programme, measured by any adverse effects to antibiotics | During the 6-month follow-up.
  The tolerance level to the Weekly Oral Cyclic Antibiotic Programme, measured by any adverse effects to antibiotics
The global antibiotic consumption. | During the 6-month follow-up
  The global antibiotic consumption.
The number of urine culture negative | During the 6-month follow-up
  The number of urine culture negative
The emergence of multi-resistant bacteria in urine (cultures), digestive bacteria (anal swabs), oro-pharynx bacteria (nasal swabs), and semi-quantitative research of multi-resistant bacteria in the stool. | During the 6-month follow-up
  The emergence of multi-resistant bacteria in urine (cultures), digestive bacteria (anal swabs), oro-pharynx bacteria (nasal swabs), and semi-quantitative research of multi-resistant bacteria in the stool.
the quality of life | During the 6-month follow-up
  A scale to measure the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Louis BERNARD, MD-PhD, Principal Investigator — University Hospital, Tours
Locations (4):
- France (4):
  - University Hospital, Raymond Poincaré / APHP, Garches
  - University Hospital, St Jacques / NANTES, Nantes
  - University Hospital, Pontchaillou / RENNES, Rennes
  - University Hospital, Bretonneau / TOURS, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dinh A, Hallouin-Bernard MC, Davido B, Lemaignen A, Bouchand F, Duran C, Even A, Denys P, Perrouin-Verbe B, Sotto A, Lavigne JP, Bruyere F, Grall N, Tavernier E, Bernard L. Weekly Sequential Antibioprophylaxis for Recurrent Urinary Tract Infections Among Patients With Neurogenic Bladder: A Randomized Controlled Trial. Clin Infect Dis. 2020 Dec 15;71(12):3128-3135. doi: 10.1093/cid/ciz1207. PMID 31867616